CLINICAL TRIAL: NCT02257879
Title: A Pharmacokinetic Study to Assess and Compare the Drug Interaction Risk of the Grapefruit Juice and Dietary Supplements Known to Inhibit CYP3A Enzyme Activity
Brief Title: DHB Supplement Interaction Study
Status: Withdrawn | Type: Observational
Why Stopped: due to constraints with collaborator and subject matter expert, recruitment was unable to begin
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140204; 14-E-0204
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
Keywords: Midazolam; CYP3A; Loperamide

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Sequence A: water - GFJ - supplement
- Sequence B: GFJ - supplement - water
- Sequence C: supplement - water - GFJ

SUMMARY:
Background:

- Drinking grapefruit juice changes how long it takes some medicines to be broken down in the body. Researchers have found that a substance in grapefruit juice called DHB contributes to this effect. Some dietary supplements contain DHB and claim to increase the absorption of any and all supplements, medicine or any other drug. But these usually contain a lot more DHB than a glass of grapefruit juice. Researchers want to study the effects of grapefruit juice and supplements with DHB.

Objective:

- To compare how a certain dietary supplement (sold as DHB-300 ) versus grapefruit juice affects how long it takes a person s body to break down medicines.

Eligibility:

- Healthy volunteers ages 18 - 60.

Design:

* Participants will be screened with medical history, physical exam, and blood and urine tests.
* Participants will have 3 treatment visits. Participants cannot drive themselves home from the visits. Each visit lasts about 13.5 hours and includes:
* Questions about medications and participant s health.
* Vital signs taken.
* A finger probe to measure oxygen.
* Blood and urine sampling throughout the visit.
* An IV line inserted into an arm vein. It will stay there throughout the visit.
* Study treatments:
* Midazolam hydrochloride a syrup given to make people sleepy.
* Loperamide a tablet for treating diarrhea.
* 1 glass of water, 1 glass of grapefruit juice, or 1 pill of DHB-300. A different one will be given at each treatment visit.
* One week before each visit, participants cannot have certain fruits and juices. They must fast the night before each visit.
* For the 3 days after each visit, participants will return to the clinic 4 times. Their vital signs will be checked and blood will be drawn.

DETAILED DESCRIPTION:
6 ,7 -dihydroxybergamottin (DHB) is one of the components of grapefruit juice and is a known irreversible inhibitor of intestinal cytochrome P450 3A (CYP3A). A single serving (240 mL) of grapefruit juice (GFJ) contains less than or equal to 5 mg of DHB. The pharmacokinetic boosting effect of GFJ has fueled the marketing of dietary supplements labeled to contain DHB e.g. DHB 300 (TM) and Trisorbagen that enhance absorption naturally, While these supplements have been found to inhibit CYP3A activity, the DHB content in these supplements is much lower than that, of GFJ. Moreover, the effects of such supplements on the pharmacokinetics of CYP3A-metabolized drugs are largely unknown. This single-center, open-label, randomized, 3-period, single-dose, crossover study in healthy volunteers will compare the drug interaction risk of a dietary supplement known to affect CYP3A with GFJ. The primary objective of this study is to compare the effects of a supplement known to affect CYP3A (e.g.Trisorbagen) with those of GFJ and water on the pharmacokinetics of two model substrates, the FDA-recommended CYP3A probe substrate midazolam, and the dual CYP3A/P-glycoprotein (P-gp) substrate loperamide. This dual-probe substrate approach to assess drug interaction risk will provide mechanistic insight into any interaction observed. Eligible volunteers (n=12) will undergo 3 phases, each comprising an exposure visit and 4 subsequent post-exposure visits to collect blood and urine over 72 or 12 hours, respectively. Exposure visits will be scheduled at least 2 weeks apart to allow washout between the phases. At each exposure visit, participants will be administered oral doses of midazolam hydrochloride (2.5 mg) and loperamide (16 mg) concomitantly with water (240 mL), GFJ (240 mL), or Trisorbagen (with 240 mL water) according to a randomized treatment sequence. Blood and urine will be collected pre-dose and post-dose over 72 (blood) or 12 (urine) hours for subsequent analyses of relevant pharmacokinetic outcomes of each probe substrate, including the primary endpoints area under the concentration-time curve from time zero (pre-dose) to infinity (AUC0-inf) and maximum observed concentration (Cmax). Secondary endpoints include geometric means, estimates of treatment differences, within-subject and between-subject treatment variance, as well as the 95% confidence intervals around those estimates.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-60
* Men and non-pregnant women
* Participant in the Environmental Polymorphisms Registry. Prior to enrollment in this study the participant will be required to enroll in the -Environmental Polymorphisms Registry.
* Willing to abstain from fruit juices, star fruit, grapefruit and grapefruit-related fruits (e.g., pomelo, Seville orange), and grapefruitcontaining products for 1 week prior to Exposure Visits and for the 4 follow-up visits.
* Willing to fast (with the exception of water) from midnight prior to the screening visit and each Exposure Visit, including abstaining from

alcohol and caffeinated beverages

-Ability to successfully complete treatment visits, including securing transportation

EXCLUSION CRITERIA:

* Women who are currently pregnant or breastfeeding
* Current use of known CYP3A inhibitors or inducers, which in the opinion of the Investigator poses an unacceptable risk to the patient or to the validity of study results. Candidates will be asked about medication use during the screening process and on the day of the exposure visits. The collected data will be reviewed by the PI or designee to confirm the candidates eligibility.
* Known liver dysfunction or disease as defined by:

  * ALT - higher than the normative value and/or determined abnormal by the PI
  * AST higher than the normative value and/or determined abnormal by the PI
  * ALP higher than the normative value and/or determined abnormal by the PI

Known kidney dysfunction or disease or:

* Estimated Glomerular Filtration Rate (eGFR)- <60 ml/min per the MDRD equation

  * Heart disease
  * Pre-existing and known history of psychiatric disorders
  * Known history of Myasthenia gravis
  * Current use of quinidine, ritonavir, and saquinavir (potential interaction with loperamide)
  * Current use of study drug-related medications (benzodiazepines, opioids, herbal supplements; temporary discontinuation per the investigator s discretion may be allowed). Candidates will be asked about medication use during the screening process and also during each of their exposure visits. The collected data will be reviewed by the PI or designee to confirm the candidates eligibility.
  * Known allergy or hypersensitivity to any study treatments (i.e., to GFJ, DHB, midazolam, loperamide, green, black or white pepper, and -Indian Gooseberry),any opioids, or benzodiazepines
  * History of acute-angle glaucoma
  * History of sleep apnea
  * Current diagnosis of anemia, as defined by hemoglobin concentration <13 g/dL for males and hemoglobin concentration <11 g/dL for females or hematocrit values (determined by lancet-induced drop of blood from the fingertip or via clinical labs) Hematocrit must be at least 34% for women and 36% for men on every visit.
  * Blood donation within the past 8 weeks of the exposure visit.
  * Use of medications for which consumption of GFJ is contraindicated and which in the opinion of the Investigator would pose an unacceptable risk to the patient if discontinued or continued while consuming GFJ. Candidates will be asked about medication use during the screening process. The collected data will be reviewed by the PI or designee to confirm the candidates eligibility.
  * Any other conditions or substance use that in the opinion of the Investigator would pose an unacceptable risk to the patient or to the validity of the study results. Candidates will be asked about health conditions during the screening process. The collected data will be reviewed by the PI or designee to confirm the candidates eligibility.
  * BMI >35.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the Environmental Polymorphisms Registry. Prior to enrollment in this study the participant will be required to enroll in the Environmental Polymorphisms Registry.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measures (AUC0 inf, Cmax) of systemic drug exposure | AUC from 0-72 h -inf
  PK measures of systemic probe drug exposure (AUCO-inf and Cmax), determined via conventional non-compartmental methods using Phoenix WinNonlin (v6.2)

SECONDARY OUTCOMES:
Geometric means, estimates of treatment differences, within-subject and between-subject treatment variance, and the 95% confidence intervals around those estimates | AUC from 0-72 h -inf

CONTACTS AND LOCATIONS:
Overall Officials: Shepherd H Schurman, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] de Castro WV, Mertens-Talcott S, Derendorf H, Butterweck V. Grapefruit juice-drug interactions: Grapefruit juice and its components inhibit P-glycoprotein (ABCB1) mediated transport of talinolol in Caco-2 cells. J Pharm Sci. 2007 Oct;96(10):2808-17. doi: 10.1002/jps.20975. PMID 17542018
- [Background] Paine MF, Oberlies NH. Clinical relevance of the small intestine as an organ of drug elimination: drug-fruit juice interactions. Expert Opin Drug Metab Toxicol. 2007 Feb;3(1):67-80. doi: 10.1517/17425255.3.1.67. PMID 17269895
- [Background] Lang M, Seifert MH, Wolf KK, Aschenbrenner A, Baumgartner R, Wieber T, Trentinaglia V, Blisse M, Tajima N, Yamashita T, Vitt D, Noda H. Discovery and hit-to-lead optimization of novel allosteric glucokinase activators. Bioorg Med Chem Lett. 2011 Sep 15;21(18):5417-22. doi: 10.1016/j.bmcl.2011.06.128. Epub 2011 Jul 18. PMID 21813277
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-E-0204.html